CLINICAL TRIAL: NCT06596434
Title: 4-Aminopyridine to Treat Skin Burns
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: John Elfar (Other)
Responsible Party: Sponsor-Investigator, John Elfar, Tenured Professor, Chairman, Department of Orthopaedic Surgery, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00005193
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Burns; Second Degree Burn; Wounds and Injuries
Keywords: 4-aminopyridine; 4-AP; Burns; Second degree burn; Wounds
MeSH Terms: conditions — Burns; Wounds and Injuries | interventions — 4-Aminopyridine

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, placebo-controlled trial design.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects in both aims will be assigned to Group A or Group B using a randomization scheme. Each study participant for each aim is randomly assigned to either treatment or placebo using permuted block randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: 4-aminopyridine (Active Comparator): Dalfampridine (generic) 10 mg capsule PO every 12 hours
  Interventions: Drug: Drug: 4-Aminopyridine
- Group B: Placebo (Placebo Comparator): Placebo - 1 capsule PO every 12 hours
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Drug: 4-Aminopyridine — Active study drug
  Other Names: 4AP; 4-AP; Dalfampridine
  Arms: Group A: 4-aminopyridine
Other: Placebo — Placebo comparator
  Arms: Group B: Placebo

SUMMARY:
Many patients suffer from traumatic burns and current treatments do not increase the regenerative potential of either skin grafts or the remaining uninjured skin. There is a need to develop treatments to accelerate and improve healing of burn injuries. More research is needed to evaluate the role of 4-AP, a promising new agent with an excellent safety profile, on wound and burn healing. The investigational treatment will be used to test the hypothesis that 4-AP accelerates burn healing in traumatically burned patients.

DETAILED DESCRIPTION:
Burn treatment has not appreciably changed in decades. Most treatments focus on infection prevention and control, as well as fluid management. This is because burns are universally infected with bacteria allowed to infiltrate deeper tissues by the absence of a skin barrier. If bacteria can now get into these tissues, the problem is only made worse by the large amount of hydration that now can get out into the environment from the open wound. Desiccation sets in with deeper tissues losing fluids. This renders tissue significantly more susceptible to further infection, as dry tissues are less perfused and less capable of fighting infectious insults. Desiccation also robs burned patients of fluids vital to sustain cardiopulmonary function. Without skin, patients essentially lose fluids and cannot perfuse even the most vital organs with time.

Research in the field focuses on preventing complications and temporizing these two factors. No regenerative treatments are currently offered to accelerate wound healing, and few investigative treatments are ready for translation to human trials. Most of the pipelines for future treatment involve long development timelines and still focus chiefly on infection control instead of driving tissue to regenerate and heal faster. A significant gap is the need for a regenerative burn treatment that can be trialed while still allowing the use of current protocols. An adjuvant regenerative burn treatment is needed.

The purpose of this study is to evaluate the role of local 4-aminopyridine (4-AP) on the treatment of burn wounds to accelerate healing.

ELIGIBILITY:
Inclusion Criteria:

* Injured (burned) adults with a maximum severity of second-degree burns.
* Burns involving at least 6cm2 of skin area
* Acute burns within 7 days of injury
* Cognitive ability to evaluate burn healing, report sensory and motor deficit during examination.
* Adults aged 18-80
* Ability to give written informed consent.
* Capable of safely coming in for follow up visits on all scheduled appointments.

Exclusion Criteria:

* History of multiple sclerosis, stroke or any other diagnosed neurological disorder
* History of hypersensitivity to AMPYRA® or 4-aminopyridine
* Current use of aminopyridine medications, including other compounded 4-AP
* Suspected renal impairment based on the Choyke questionnaire.
* History of difficult compliance with timely follow up
* Patients outside the age range
* Unable to provide informed consent.
* Patients with a known history of a seizure disorder (4-AP overdose can, in selected cases, result in limited seizure activity).
* Patients with a concomitant traumatic brain injury.
* Patients unable to communicate.
* Patients unwilling to complete the study requirements.
* Patients currently taking organic cat-ion transporter 2 (OCT2) inhibitors, e.g. Cimetidine.
* Pregnancy, breastfeeding or incarcerated individuals.
* Non-English speaking
* Patients unable or unwilling to take calibrated (with gauge) photographs of their wounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Healing rate | 12 months
  Each subject will undergo detailed fiducial-marking augmented macroscopic imaging to determine baseline burn area measurement. These measurements will be repeated at each follow up study visit to assess healing rate.

SECONDARY OUTCOMES:
Skin-graft rate | 12 months
  Skin-graft rate (failure of healing)
Scar formation | 12 months
  Scar formation will be measured by the Patient and Observer Scar Assessment Scale (POSAS). Each item of the POSAS is rated on a 10-point score with total scores ranging from 6 to 60 with higher scores indicating increase severity of symptoms. These measurements will be repeated at each follow up study visit.
Scar sensitivity | 12 months
  Scar sensitivity will be measured by the Patient and Observer Scar Assessment Scale (POSAS). Each item of the POSAS is rated on a 10-point score with total scores ranging from 6 to 60 with higher scores indicating increase severity of symptoms. These measurements will be repeated at each follow up study visit to assess healing rate.

CONTACTS AND LOCATIONS:
Overall Officials: John Elfar, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No